CLINICAL TRIAL: NCT06870175
Title: Non-Invasive Ambulatory Monitoring of Electrocardiogram (ECG) and Arrhythmia Detection Using Textile Electrodes
Brief Title: Smart Textile ECG Monitoring
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Myant Medical Corp. (Industry)
Collaborators: Partners in Advanced Cardiac Evaluation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5.21
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Arrhythmia
Keywords: Smart Textile; Ambulatory Electrocardiogram Monitoring; Holter Monitoring; Arrhythmia detection; Textile electrodes
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adults with cardiovascular disease and/or risk factors (Experimental): In this study, a total of 300 participants are expected to participate, specifically: The target population for this study are adults above 18 years of age with cardiovascular disease and/or risk factors, who have been prescribed a 14-day ambulatory ECG monitoring by their physician.
  Interventions: Device: Electronic-Textile-based Electrocardiographic Monitoring

INTERVENTIONS:
Device: Electronic-Textile-based Electrocardiographic Monitoring — Participants will be invited to wear the Skiin chest band for up to 14 days, as prescribed by their physician. Participants will wear the Skiin chest band in a similar capacity to a conventional Holter monitor.

SUMMARY:
This research is a clinical evaluation of the Skiin chest band, a smart garment with embedded electronic textile (e-textile) electrodes, to record body surface electrocardiogram (ECG) signals. Developed by Myant Textile Computing Inc., the Skiin chest band (i.e. as part of the Skiin Underwear family of garments) is a component of the Myant Health Platform (MHP). The MHP also consists of: (a) a mobile phone application (Skiin Connected Life Application; SCLA), and (b) the Myant Virtual Clinic Portal (MVCP). In this study, participants will wear the Skiin chest band to collect their ECG for a period of 14 days. Participants will also be provided with a smartphone that is pre-loaded with the SCLA to record any symptoms (e.g. palpitations, shortness of breath, fatigue, light- headedness, fainting, etc.) they may experience over the 14 day ECG monitoring period. The data collected in this study will be used to develop new algorithms and patient monitoring tools to detect and predict cardiovascular health problems.

ELIGIBILITY:
Inclusion Criteria:

* Being referred to the Partners in Advanced Cardiac Evaluation (PACE Cardiology), and having been prescribed a 14-day ambulatory ECG monitoring by their physician.
* Able to understand and speak English language, enough to provide informed consent.

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Cardiovascular Implantable Electronic Devices (CIED), including Implanted cardioverter defibrillator (ICD) or pacemakers
* Absence of chest band that fits the participant's body
* Open wound or dressing on a body part that needs to be in contact with the Skiin garment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2026-02-19 (Estimated)

PRIMARY OUTCOMES:
Arrhythmia Detection | Each participant undergoes up to 14 day ambulatory ECG monitoring from the time of wearing the Skiin chest band.
  To evaluate the performance of Skiin chest band in collecting ambulatory body surface ECG, and in detecting the presence or absence of arrhythmias for up to 14 days

OTHER OUTCOMES:
Algorithm Validation (Arrhythmia detection) | Each participant undergoes up to 14 day ambulatory ECG monitoring from the time of wearing the Skiin chest band.
  To validate an artificial intelligence/ machine learning (AI/ML) arrhythmia detection algorithm
Algorithm Validation (Atrial Fibrillation Burden) | Each participant undergoes up to 14 day ambulatory ECG monitoring from the time of wearing the Skiin chest band.
  To use the AI/ML arrhythmia detection algorithm to establish Atrial Fibrillation burden, defined as: the ratio of time spent in Atrial Fibrillation over total monitoring duration (i.e. up to 14 days)
Usability Rating | Each participant undergoes up to 14 day ambulatory ECG monitoring from the time of wearing the Skiin chest band.
  To evaluate the usability of the Skiin chest band for ambulatory ECG monitoring, as rated by study participants on the associated usability questionnaire. The questionnaire, entitled "Smart Textile ECG Monitoring (PACE-MYANT) - Usability Questionnaire". The questionnaire includes 16 questions that are answered on a 7-point Likert scale, in addition to other questions, where participants.
  The ratings in the the 7-point Likert scale (sections A) are "Strongly Disagree", "Disagree", Somewhat Disagree", "Neither agree nor disagree", "Somewhat Agree", "Agree", "Strongly Agree". Higher ratings and scores indicate better usability and overall experience.
  The ratings in the sections C are from 1 to 7: "Strongly favor other Holter", "Favor other Holter", "Somewhat Favor other Holter", "No preference", "Somewhat favor Skiin", "Favor Skiin", "Strongly favor Skiin". Higher ratings and scores indicate preference for Skiin vs. standard Holter monitoring with wires and adhesive patches.
Clinic Workflow Statistics | Before and after ambulatory ECG monitoring (up to 14 days) for each patient
  To document workflow statistics for Skiin ambulatory ECG monitoring in terms of (a) patient set-up s (i.e. the time it takes (in minutes) to set up a patient with the Skiin, and (b) report processing time (i.e. the time it takes for the ECG technician to scan/process the ambulatory ECG results?

CONTACTS AND LOCATIONS:
Overall Officials: Mouhannad Sadek, MD, Principal Investigator — Partners in Advanced Cardiac Evaluation (PACE)
Locations (1):
- Partners in Advanced Cardiac Evaluation (PACE) Cardiology Clinic, Newmarket, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No